CLINICAL TRIAL: NCT00163345
Title: Evaluation of Parameters of the Small Airways and Their Changes Under Treatment With Ciclesonide (320 mcg Once Daily) Versus Placebo in Patients With Asthma
Brief Title: Efficacy of Ciclesonide on Small Airways in Patients With Stable Asthma (18 to 60 y) (BY9010/M1-131)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY9010/M1-131
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Asthma
Keywords: Asthma; Ciclesonide; Small Airways
MeSH Terms: conditions — Asthma | interventions — ciclesonide

INTERVENTIONS:
Drug: Ciclesonide

SUMMARY:
The aim of this study is to evaluate the involvement of small airways in asthma, as determined by bronchial challenges, CT-scanning, and cellular markers of inflammation. Ciclesonide will be inhaled at one dose level once daily. The study duration consists of a baseline period (2 to 3 weeks) and a treatment period (5 to 6 weeks). The study will provide further data on safety and tolerability of ciclesonide.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent
* History of bronchial asthma
* FEV1 more than or equal to 60% of predicted
* Stable asthma
* Patients who are in good health with the exception of asthma

Main Exclusion Criteria:

* Concomitant severe diseases, diseases expected to interfere with the outcome of the study, or diseases which are contraindications for the use of ICS
* COPD (i.e. chronic bronchitis or emphysema) and/or other relevant lung diseases causing alternating impairment in lung function
* Use of ICS 4 weeks before entry into the baseline period
* Pregnancy
* Intention to become pregnant during the course of the study
* Breast feeding
* Lack of safe contraception
* Use of other drugs not allowed
* Current smokers and ex-smokers with more than or equal to 10 pack-years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2003-09; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
variables of primary interest are FVC% at PC20 MCh, SVC% at PC20 MCh
FVC% at PC20 AMP, SVC% at PC20 AMP
regional air trapping
bronchial and alveolar exhaled NO
lung function variables
non-cellular inflammatory markers.

SECONDARY OUTCOMES:
safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- Altana Pharma/Nycomed, RB Groningen, Netherlands

REFERENCES:
- [Derived] Cohen J, Douma WR, ten Hacken NH, Vonk JM, Oudkerk M, Postma DS. Ciclesonide improves measures of small airway involvement in asthma. Eur Respir J. 2008 Jun;31(6):1213-20. doi: 10.1183/09031936.00082407. Epub 2008 Feb 20. PMID 18287130
- See also: BY9010_M1-131 Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4498&filename=BY9010_M1-131%20Synopsis.AZCT.com%20posting.pdf